CLINICAL TRIAL: NCT02908971
Title: Association Between Soy Based Formula Consumption During Infancy and the Timing of Pubertal Signs and BMI-SDS
Brief Title: Association Between Soy Based Formula in Infancy and Puberty
Status: Completed | Type: Observational
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Assaf harofeh Medical Center, Assaf-Harofeh Medical Center
Other Study IDs: 257/15
Record Dates: First submitted 2016-09-18; First posted 2016-09-21 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Puberty and Body Composition
Keywords: soy based formula; overweight; adrenarche,; gonadarache
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Soy based formula: "soy group" will include children from the children who had milk allergy, and consumed a soy-based substitute formula for longer than three months and agreed to participate in this study.
  Interventions: Behavioral: soy based formula at infancy
- Healthy control: The control group will included children (at a rate of 2:1) who will be assigned randomly from the healthy population at the initial cohort, and who will agree to participate.

INTERVENTIONS:
Behavioral: soy based formula at infancy — The intervention is only past history of soy consumption
  Groups: Soy based formula

SUMMARY:
Background: Children in industrialized and developing countries have a higher tendency to present earlier signs of puberty. One hypothesis includes the hormonal effects of phytoestrogens found in soy products.

Objective: to examine the association between consumption of soy-based food in early infancy and childhood and the incidence of early or precocious puberty and overweight in school-aged children.

Methods: the study population for this case control study is randomized from a prospectively followed cohort of all babies born at Assaf Haroffeh medical center and followed for milk allergy signs and food intake until the age of 3 years (A nested cohort). It is divided to those who were allergic to milk, and thus consumed only soy based formula and food during infancy and childhood (soy group) and a randomized control group who consumed non-soy based intake. For both groups data are available of food habits during infancy and collected from 3 days food diaries during the current study. Physical examination, including weight , height, blood pressure and Tanner Pubertal Staging will performed annually.

DETAILED DESCRIPTION:
Soy and soy-based products are widely used in modern day nutrition. It is widely consumed among all populations, especially among vegetarians, vegans, those with milk allergy, and in the general population who consume processed foods .Soy-based infant formula is commonly used, and may account for nearly 25 % of the infant formula sold . Soy products contain phytoestrogens (isoflavones) that were suggested to function as weak hormonal disruptors due to their functional similarity to mammalian estrogens and their active metabolites. Studies regarding the effects of soy consumption on pediatric growth and body mass have been inconclusive. Infants who are fed soy-based formulas have higher isoflavones blood concentration compared to breast-fed and milk-based formulas fed babies . Several studies discuss its effect on infantile physiologic telarche . Several retrospective, case-control and case studies were reported trying to elucidate the possible clinical association between consumption of soy products during infancy and childhood and pubertal and menarchal timing. However, there results are contradictory and inconclusive .Furthermore, in some of the studies there is no discussion of the association or confounding effect of overweight which is also associated with pubertal timing. Despite the importance of the topic, there is paucity of prospective data regarding the impact of soy based products consumption on puberty and body mass index (BMI).

Thus, this prospective study will examine the relationship between the consumption of soy- based formulas in early infancy with the development of early puberty and changes in anthropometric measures in school-aged children. The goal of this study is to test the association between early consumption of soy based formula and the timing of onset of secondary sexual characteristics in a prospective mannor and with consideration of current dietary intake and confounding factors as BMI and familial trends.

MATERIALS AND METHODS Study Population The study population is based on a large cohort study initiated and performed during 2004-2006 by Katz Y et al ,which followed prospectively all newborns born during this time period at Assaf Haroffeh Medical Center, Zerifin, Israel.The study looked into their nutritional intake, development of sensitivity to milk and milk allergies. The population included a total of 13019 children, out of which 66 developed an IgE-mediated Cow Milk Allergy (CMA), 71 developed milk-sensitivity, and 12638 were healthy. Our study population includes all CMA group and a randomized group from the healthy population (nested cohort).

Inclusion criteria : all participants from initial study . Exclusion criteria:lack of data regarding food intake during infancy in both groups. In the non-allergic children, from the non soy based group those who consumed soy - based formula for religious or ideological reasons will be excluded.

Study design This is a case-control study, including a specific sub-population from a large cohort population including prospectively collected data on infantile food consumption. All original cohort participants, who fulfill the inclusion criteria will be approached for participation in the current study. The current study will include demographic and clinical data collection, an interview and 3 days of food diary preparation and dietician analysis and a physical examination by a pediatric Endocrinologist.

Demographic and clinical data Collection Data will include the information from the initial prospective follow up at infancy including birth weight, birth week, parental origin, infantile food habits, maternal age and allergy classification. Data collected at the current session: family health history including obesity, early or delayed puberty, ,age of maternal menarche and age of paternal shaving, parental height. The child physical activity levels and nutritional habits, illnesses, medications . Height and weight were measured and body mass index [BMI] will calculated and reported as BMI-SDS . Tanner score was used to characterize sexual maturation. The pre-pubertal state was defined as Tanner stage 1 genitalia and testicular volume ≤3 ml in boys and absence of breast development in girls. A specific description of axillary odor and axillary hair and pubertal hair will be performed for adrenarche signs.

Dietary intake analysis All participants will fill a detailed 3 days food diary (two weekdays and one weekend day) according to guidance by the study dietician. The nutritional data from the food records will be analyzed using the Tzameret Program (or A computer program, based on local food tables, developed by Israeli ministry of Health) ).Results of the analysis will be reported as percent-Dietary Reference Intakes (DRI).

ELIGIBILITY:
Inclusion Criteria: All participants of initial cohort of children born 2004-2006 -

Exclusion Criteria: Those from soy group who did not consume soy based formula. Those from healthy control who did consume soy formula.

Refusal for physical examination.

-

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study population is based on a large cohort study initiated and performed during 2004-2006 by Katz Y et al , which followed prospectively all newborns born during this time period at Assaf Haroffeh Medical Center, Zerifin, Israel . The study looked into their nutritional intake, development of sensitivity to milk and milk allergies. The population included a total of 13019 children, out of which 66 developed an IgE-mediated Cow Milk Allergy (CMA), 71 developed milk-sensitivity, and 12638 were healthy. Our study population included all CMA group and a randomized group from the healthy population (nested cohort).
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Age of adrenarche signs | 5 years
  Age of adrenarche signs will be compared between soy and control groups
Age of gonadarche signs | 5 years
  Age of gonadarche signs will be compared between soy and control groups

SECONDARY OUTCOMES:
comparison of rate of Overweight and obesity | 5 years
  BMI-SDS will be compared between groups

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Rachmiel, MD, Principal Investigator — Assaf Haroffeh Medical Center
Locations (1):
- Assaf Haroffeh Medical center, Ẕerifin, Israel

IPD SHARING:
Plan to Share IPD: No